CLINICAL TRIAL: NCT05513404
Title: Acute Study of Polyphenol-rich Honeyberries, Cherries, and Raspberries Grown in Scotland on Postprandial Glycaemic Response
Brief Title: The Scottish Fruit Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2022_01/ROW-Honeyberry
Record Dates: First submitted 2022-08-19; First posted 2022-08-24 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Postprandial Hypoglycemia; Age-Related Memory Disorders
Keywords: blood glucose; acute glycemic response; postprandial glycemia; short term memory; soft fruits; honeyberry; raspberry; cherry
MeSH Terms: conditions — Hypoglycemia; Memory Disorders

STUDY DESIGN:
Intervention Model Description: This acute intervention study will have a randomised controlled crossover design where the volunteers will return for 4 stand-alone study sessions. All study procedures will be carried out at the Human Nutrition Unit (HNU) of the Rowett Institute.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Breakfast only (No Intervention): This is an acute intervention study to compare the health benefits, in relation to changes in postprandial glucose and cognitive performance, of consumption of 3 soft fruits, raspberries, cherries, and honeyberries. It will have a randomised controlled crossover design where the volunteers will return for 4 stand-alone study sessions. All study procedures will be carried out at the Human Nutrition Unit (HNU) of the Rowett Institute. . The first study session will be an oral glucose tolerance test (OGTT). The glucose load for the OGTT in all sessions will be given as carbohydrate meal consisting of white bread, spread, low-polyphenol jam. (meal: 75g carbohydrate total). The remaining three will be intervention sessions which will be identical in all respects except for the addition of either honeyberry, cherry, or raspberry. There will be a minimum of 1 week washout period.
- Honeyberry (Experimental): This arm will be an oral glucose tolerance test (OGTT). The glucose load for the OGTT in all sessions will be given as carbohydrate meal consisting of white bread, spread, low-polyphenol jam. (meal: 75g carbohydrate total) with the addition of honeyberry. There will be a minimum of 1 week washout period.
  Interventions: Dietary Supplement: Honeyberry
- Cherry (Experimental): This arm will be an oral glucose tolerance test (OGTT). The glucose load for the OGTT in all sessions will be given as carbohydrate meal consisting of white bread, spread, low-polyphenol jam. (meal: 75g carbohydrate total) with the addition of cherrry. There will be a minimum of 1 week washout period.
  Interventions: Dietary Supplement: Cherry
- Raspberry (Experimental): This arm will be an oral glucose tolerance test (OGTT). The glucose load for the OGTT in all sessions will be given as carbohydrate meal consisting of white bread, spread, low-polyphenol jam. (meal: 75g carbohydrate total) with the addition of raspberry. There will be a minimum of 1 week washout period.
  Interventions: Dietary Supplement: Raspberry

INTERVENTIONS:
Dietary Supplement: Honeyberry — To investigate changes in postprandial glucose and cognitive performance, after consumption of honeyberries grown in Scotland.
  Arms: Honeyberry
Dietary Supplement: Cherry — To investigate changes in postprandial glucose and cognitive performance, after consumption of cherries grown in Scotland.
  Arms: Cherry
Dietary Supplement: Raspberry — To investigate changes in postprandial glucose and cognitive performance, after consumption of raspberries grown in Scotland.
  Arms: Raspberry

SUMMARY:
The purpose of this study is to determine if new varieties of fruits grown in Scotland which can adapt better to climate change namely, honeyberries and cherries, have the same health benefits as established fruits such as raspberries. To do this we will investigate the effects of consuming honeyberries, cherries, and raspberries on short term changes in blood glucose, and on short term memory.

DETAILED DESCRIPTION:
As humans spend most of their day in a postprandial state, it is imperative that the metabolic effects of diets are well understood if the incidence of chronic disorders such as type 2 diabetes (T2D) is to be controlled. Current estimates place global incidence of diabetes at 537 million, and this number is predicted to rise a further 45% by 2045. T2D is linked to increased risk of developing other chronic health conditions including cardiovascular disease (CVD) and dementia.

Controlling the acute glycaemic response and avoiding hyperglycaemia is essential for reducing diabetic risk. In addition, acute hyperglycaemia may provoke metabolic reactions increasing CVD risk and lower episodic memory even in non-diabetic individuals. Diet has an important role to play, and modern Western diets typically have high glycaemic loads due to excessive refined and total carbohydrate contents. As a result, the average blood glucose concentration of individuals has increased over the past three decades.

Polyphenolic constituents of foods may help to delay starch and disaccharide digestion and glucose absorption following a carbohydrate-containing meal or beverage. In vitro studies suggest that some polyphenols found in fruits are effective inhibitors of digestive enzymes, α-amylases and α-glucosidases and inhibit the action of intestinal glucose transporters. There is only a small amount of information available from human studies however, randomized controlled trials (RCTs) have shown that fruits reduced postprandial glucose concentrations following consumption of either starch, glucose or sucrose loads. Strategies to control chronic postprandial hyperglycaemia through increased consumption of such polyphenol rich foods would strengthen efforts to reduce the risk of developing T2D in the general population.

The aim of this study is to test the health benefits of new climate resistant fruit high in polyphenols grown in Scotland with and an existing crop already established in the fruit market. The hypothesis is that consumption of honeyberries and cherries grown in Scotland is as effective as raspberries in reducing the postprandial glycemic response in normal weight /overweight, healthy men, and post-menopausal women. With a secondary objective looking at the effects of these fruits on cognitive function.

This is a randomized cross over study and will aim to recruit 28 normal to overweight (BMI ≥ 18.5 and < 39.9), men or post-menopausal women (post-menopausal defined as not having had a period for over a year), aged ≥40 and ≤ 70 years who will attend four study sessions. The first study session will be an oral glucose tolerance test (OGTT) and the remaining three will be identical in all respects except for the addition of the fruit. Consecutive blood samples will be collected in all 4 study sessions which will be used to measure glucose, insulin, C-peptide, incretins, and lipids. Cognitive function the secondary outcome will be measured using a series of memory tests.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or post-menopausal women
* Aged ≥40 and ≤ 70 years old.
* BMI ≥ 18.5 kg/m2
* HbA1c <6.5%

Neuropsychological screening tasks will include the Mini-Mental State Examination (MMSE), the National Adult Reading Test (NART), the Geriatric Depression Scale (GDS), the Trail Making Test (TMT), the Controlled Oral Word Association Test (COWAT), the Hopkins Verbal Learning Test (HVLT),

* MMSE >= 27
* NART, TMT, COWAT and HVLT within acceptable norms

Exclusion Criteria:

* Exclusion Criteria

Those with any of the following will be excluded from participation:

We will ask the volunteers to complete a questionnaire to state current health complaints and current medication use.

Chronic illness, including: thromboembolic or coagulation disease unregulated thyroid disease kidney disease hepatic disease severe gastrointestinal disorders pulmonary disease (e.g. chronic bronchitis, COPD, pacemaker implant) Alcohol or any other substance abuse Eating disorders a history of neurological abnormalities, Women who are lactating or breastfeeding, pregnant Allergic/intolerant to foods provided in the study (Fruit allergy). Alcohol and/or other substance abuse Smoking and the use of e-cigarettes Physically active at a competitive level (exercising strenuously on a daily basis for long periods of time)

Medication exclusion criteria Oral steroids Tricyclic antidepressants, neuroleptics Anticoagulants Digoxin and anti-arrhythmics Insulin, Sulphonylureas, Thiazolidinediones (glitazones), metformin. Chronic use of anti-inflammatories (e.g. > 200mgs doses of aspirin, ibuprofen), current psycho-active medication chlorphenamine

Neuropsychological exclusion criteria

* MMSE < 27
* GDS > 5
* Self-report of prior diagnosis of dementia, probable dementia, or mild cognitive impairment
* History of stroke, severe head injury or other neurological condition which may adversely affect cognition
* history of anxiety and depression

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in postprandial glucose response associated with glycaemia in healthy normal/overweight men and post-menopausal women (40-70 years) when honeyberries, cherries or raspberries grown in Scotland are ingested. | 4 hours
  Based on our previous studies assuming a within-person spread of 10% (as observed previously), 16 volunteers are needed to detect a change in postprandial glucose response of 12% or more, with a power of 80% at the 5% significance level which is the primary outcome.
Change from baseline in postprandial episodic memory in healthy normal/overweight men and post-menopausal women (40-70 years) when honeyberries, cherries or raspberries grown in Scotland are ingested. | 4 hours
  From a previous study on honeyberry and assuming a within-person variability for the episodic memory tests of 1.92, to detect a change in episodic memory of 15% requires 28 volunteers for 80% power.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona M Campbell, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- Rowett Research Institute, University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No